CLINICAL TRIAL: NCT04635384
Title: Assessment of Chimerism and Relapse Post Bone Marrow/HCT Transplant Using AlloHeme Test (ACROBAT)
Brief Title: Assessment of Chimerism and Relapse Post Bone Marrow/Hematopoietic Cell Transplant (HCT) Using AlloHeme Test
Acronym: ACROBAT
Status: Active, not recruiting | Type: Observational
Sponsor: CareDx (Industry)
Responsible Party: Sponsor
Other Study IDs: SN-C-00014
Record Dates: First submitted 2020-10-28; First posted 2020-11-19 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2024-10

CONDITIONS: Acute Myeloid Leukemia; Acute Lymphoblastic Leukemia; Myelodysplastic Syndrome
Keywords: AML; ALL; MDS
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Myelodysplastic Syndromes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — AlloHeme is a chimerism test service that utilizes NGS technology to analyze SNP loci to quantify donor and recipient cells by measuring genomic DNA. Before transplant, patient and donor peripheral blood sample will be collected to identify informative marker for routine chimerism testing and baseline establishment for AlloHeme. Post-transplant blood or bone marrow samples are obtained and compared to the baseline sample profiles to calculate % chimerism of recipient cells in the blood and/or bone marrow samples.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
AlloHeme is a chimerism test service that utilizes NGS technology to analyze SNP loci to quantify donor and recipient cells by measuring genomic DNA. Before transplant, patient and donor peripheral blood sample will be collected to identify informative marker for routine chimerism testing and baseline establishment for AlloHeme. Post-transplant blood or bone marrow samples are obtained and compared to the baseline sample profiles to calculate % chimerism of recipient cells in the blood and/or bone marrow samples. Cell selection from blood and bone marrow samples is applied to evaluate chimerism in specific cell subtypes that are relevant to AML and MDS diseases (CD3+ T lymphocytes, CD33+ Myeloid cells and CD15+ Granulocyte cell subtypes from blood and CD34+ hematopoietic stem cells from bone marrow).

DETAILED DESCRIPTION:
The test will be started from month 1 post HCT and will be performed bi-weekly up to month 3, monthly from month 4-6 and quarterly from month 9 to year 2 for total 15 visits. During each visit, about 18 ml (3.6 teaspoons) of whole blood will be collected into 3 pink BD Hemogard tubes with K2 EDTA additive. In addition to blood collection, the subject will be asked to provide 3ml or 0.6 teaspoon of bone marrow specimens during the routine visits on Day 100(month 3), Day 180 and Day 360 for use in this research study. When bone marrow study is performed, marrow specimen will be collected for AlloHeme test at central lab. Standard chimerism assessment, bone marrow study and MRD test will be performed at each participated institution lab as clinically indicated and based on treating physician's discretion. Method of standard of care chimerism and MRD assessment will be based on each institutional standard protocol. Data related to AlloHeme test, clinical outcomes, PHI and all standard of care of patient management information will be collected from medical records. During the Baseline and pre transplant the following clinical data will be collected: sex, age, donor and recipient demographic, chemotherapy, remission status pre-transplant, donor type, HLA, stem cell source, conditioning regimen type and intensity, cytogenetics test, minimal residual disease, chimerism, T cell depletion and GVHD protocol. Following transplantation, clinical events including death, relapse, second allo-HSCT, DLI as well as the events that impact the chimerism like tapering IST, GVHD and infection will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged 18 years or above.
* The patient must have one of the following diseases: AML, ALL or MDS
* Eligible for allogeneic hematopoietic stem cell transplant
* Subjects must receive an Allo-HCT from an HLA matched related or unrelated donor or haploidentical donor
* Myeloablative or reduced intensity/non-myeloablative conditioning
* Any GVHD prophylaxis regimen including post-transplantation cyclophosphamide-based or conventional regimen
* The subject must be enrolled prior to Allo-HCT

Exclusion Criteria:

The participant may not enter the study if ANY of the following apply:

* Has history of prior Allo-HCT
* T cell depleted transplant (Including in vivo and ex vivo T cell depletion)
* Inability to comply with medical recommendations or follow-up
* Donor is identical twin
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants aged > 18 years old with a diagnosis of AML, ALL, and MDS who will undergo an Allo-HCT will be invited to participate and enrolled into the study at the time initial transplant evaluation or at any time before admission for transplantation.
Sampling Method: Probability Sample
Enrollment: 307 (Actual)
Dates: Start 2021-06-30 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
To determine the association between increased mixed chimerism (iMC) detected by AlloHeme and post-transplant relapse in patients with acute leukemia and myelodysplastic syndrome. | Jan-2022
  Comparison of cumulative incidence of relapse post-transplant of patients with increased mixed chimerism (iMC) vs. complete chimerism (CC) vs. stable/decrease mixed chimerism (sMC/dMC) detected by AlloHeme.

SECONDARY OUTCOMES:
To determine the association of microchimerism detected by AlloHeme on post-transplant relapse in patients with acute leukemia and myelodysplastic syndrome | Jan-2022
  Comparison of cumulative incidence of relapse post-transplant of patients with microchimerism vs. CC detected by AlloHeme
To determine the association between an iMC detected by AlloHeme and disease-free survival (DFS) post-transplant in patients with acute leukemia and myelodysplastic syndrome | Jan-2022
  Comparison of DFS post-transplant in patients with iMC vs. complete chimerism (CC) vs. stable/decrease mixed chimerism (sMC/dMC) detected by AlloHeme.
To determine the correlation between peripheral blood chimerism detected by AlloHeme and post-transplant measurable residual disease (MRD) status in patients with acute leukemia and myelodysplastic syndrome | Jan-2022
  Statistical correlation and agreement of peripheral blood donor chimerism quantitatively detected by AlloHeme and post-transplant MRD from bone marrow.
To compare the performance of post-transplant chimerism measured by AlloHeme versus STR-PCR method for post-transplant relapse prediction in patients with acute leukemia and myelodysplastic syndrome. | Jan-2022
  Comparison of performance AlloHeme versus STR-PCR method for post-transplant relapse prediction including Sensitivity Specificity, Positive predictive value, negative predictive value, AuROC

CONTACTS AND LOCATIONS:
Overall Officials: Nishant Dwivedi, MD/PhD, Study Director — CareDx
Locations (10):
- United States (10):
  - University of California Irvine, Brisbane, California
  - City of Hope, Duarte, California
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Georgia Cancer Center at Augusta University, Augusta, Georgia
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Washington University in St. Louis, St Louis, Missouri
  - Columbia University Irving Medical Center, New York, New York
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - University of Utah, Salt Lake City, Utah